CLINICAL TRIAL: NCT07199595
Title: Effect of Dexmedetomidine Versus Magnesium Sulfate Infusion on Intracranial Pressure and Cerebral Perfusion Pressure in Craniotomy Using Lumbar Drain Catheter
Brief Title: Dexmedetomidine Versus Magnesium Sulfate Infusion in Craniotomy
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Hassan mostafa abdelbaky ahmed, Assistant lecturer, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: Icp
Record Dates: First submitted 2025-09-22; First posted 2025-09-30 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Craniotomy Surgery

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dexmedetomidine (Active Comparator): Dexmedetomidine: loading dose 1 µg/kg IV over 10 min after induction and then maintenance dose 0.2- 0.7 µg/kg/hr based on hemodynamic response
  Interventions: Drug: Dexamedomedine
- Mgso4 (Active Comparator): Magnesium Sulfate: Used as an IV loading dose at 20 mg/kg IV over 17 minutes as an induction agent, followed by maintenance of 10 mg/kg/h to skin closure.
  Interventions: Drug: MgSO4

INTERVENTIONS:
Drug: Dexamedomedine — Group A (the Dexmedetomidine group):
  Dexmedetomidine: loading dose 1 µg/kg IV over 10 min after induction and then maintenance dose 0.2- 0.7 µg/kg/hr based on hemodynamic response.
  Arms: Dexmedetomidine
Drug: MgSO4 — Magnesium Sulfate: Used as an IV loading dose at 20 mg/kg IV over 17 minutes as an induction agent, followed by maintenance of 10 mg/kg/h
  Arms: Mgso4

SUMMARY:
To compare the intraoperative effects of Dexmedetomidine and Magnesium Sulfate infusion on intracranial pressure and cerebral perfusion pressure in adult patients undergoing craniotomy

DETAILED DESCRIPTION:
Intracranial pressure (ICP) and cerebral perfusion pressure (CPP) are critical parameters in craniotomy patients . Effective modulation of these pressures during surgery can improve intraoperative stability and postoperative recovery . Dexmedetomidine (Dexamed) is a selective α2-adrenoceptor agonist with sedative and neuroprotective properties, known to reduce ICP without respiratory depression . Magnesium Sulfate (MgSO₄) acts as an NMDA receptor antagonist and vasodilator, promoting neuronal protection and improved cerebral blood flow . By using a lumbar drain catheter intraoperatively, direct and continuous measurement of ICP is feasible, offering real-time insight into the pharmacological effects of these agents on cerebral dynamics .

The underlying research question is as follows: Can intraoperative Dexmedetomidine as opposed to Magnesium sulfate result in better ICP and CPP management of adult craniotomy patients? Nonetheless, the individual basis of usage of Dexmedetomidine and Magnesium Sulfate in neurosurgeries has been supported by existing literature , but lack of direct comparative studies to determine the effects of the two drugs on real-time intracranial and cerebral perfusion pressure in the craniotomy . This study aims to fill the existing gap in the literature by stating the continuity of ICP monitoring with a lumbar drain, thus offering a robust and standard control environment of comparison.

Intervention Protocol

Participants will be randomly assigned to one of two groups:

Group A - Dexmedetomidine Infusion

* Loading Dose: 1 µg/kg IV over 10 minutes
* Maintenance Infusion: 0.2-0.7 µg/kg/h, titrated based on sedation level and hemodynamic response
* Infusion will carry on till skin closure.
* Monitoring: MAP, HR, ICP, CPP Group B - Magnesium Sulfate Infusion
* Loading Dose: 20 mg/kg IV over 15 minutes
* Maintenance Infusion: 10 mg/kg/h throughout the procedure
* Infusion will carry on till skin closure.
* Monitoring: MAP, HR, ICP, CPP

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65 years
* Elective craniotomy for supratentorial pathology
* No contraindication to lumbar drain insertion
* Baseline mental status is stable, allowing for a reliable postoperative neurological evaluation can be done
* ASA physical status I-III

Exclusion Criteria:

* Coagulopathy or current anticoagulation
* Severe renal or hepatic dysfunction
* Known allergy to study medications
* traumatic brain injury

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-10-20 (Estimated); Primary Completion 2026-10-01 (Estimated); Study Completion 2026-11-01 (Estimated)

PRIMARY OUTCOMES:
Change in ICP and CPP in craniotomy | o Pre-loading o After loading o Once the patient is in position (other than baseline) o After 30 min of incision (or every 30-60 min till skin closure)
  compare the intraoperative intracranial pressure (ICP) and cerebral perfusion pressure (CPP) effects of dexmedetomidine and magnesium sulfate infusion in a comparative study to determine the efficacy in adult patients undergoing craniotomy, continuous measurement was achieved with the help of a lumbar drain catheter.

IPD SHARING:
Plan to Share IPD: No